CLINICAL TRIAL: NCT00222261
Title: Aspirin Non-responsiveness and Clopidogrel Endpoint Trial.
Acronym: ASCET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Norwegian Council for Cardiovascular Diseases. (Unknown); Ada and Hagbart Waages Humanitarian and Charity Foundation (Other); Alf and Aagot Helgesens Research Foundation. (Unknown)
Responsible Party: Alf-Aage R Pettersen, MD, Ullevaal University Hospital, Oslo, Norway
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCET
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Heart Disease; Angina Pectoris; Atherosclerosis
Keywords: antiplatelet therapy; aspirin non-responders; aspirin resistance; clopidogrel; coronary heart disease; stable angina pectoris
MeSH Terms: conditions — Coronary Disease; Angina Pectoris; Atherosclerosis; Angina, Stable | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, aspirin (Active Comparator): Aspirin 160 mg
  Interventions: Drug: aspirin
- 2, clopidogrel (Active Comparator): Clopidogrel 75 mg
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: aspirin — Aspirin 160 mg once daily for two years
  Arms: 1, aspirin
Drug: clopidogrel — clopidogrel 75 mg once daily for two years
  Arms: 2, clopidogrel

SUMMARY:
In the ASCET study, 1000 patients with documented coronary heart disease will be randomized to either continued treatment with aspirin 160 mg/d or change to clopidogrel 75mg/d. Clinical endpoints will be recorded for at least 2 years and related to the initial aspirin response, assessed by the PFA-100® method, to investigate whether aspirin non-responders have higher composite event rate than responders or whether Clopidogrel treatment in patients non-responsive to aspirin will reduce their risk of future clinical events. The clinical events are the composite of unstable angina, myocardial infarction, stroke or death.

DETAILED DESCRIPTION:
Background: Aspirin is widely used as an antiplatelet drug in patients with coronary heart disease. Despite documented clinical benefit, many patients on aspirin still experience severe cardiovascular events. Several laboratory reports have shown lack of platelet inhibition in 5-40% of aspirin-treated patients, and the term aspirin resistance has been introduced. The clinical relevance of these laboratory findings is, however, still unknown. New antiplatelet drugs have been developed, and the adenosin diphosphate (ADP) receptor inhibitor clopidogrel has at least the same efficacy as aspirin with an acceptable safety profile. Laboratory methods for determination of platelet reactivity and treatment efficacy have been complicated and time consuming. New methodologies, like the PFA-100® system, have made such analyses more suitable for clinical use.

Design: In the ASCET study, 1000 patients with documented coronary heart disease will be randomized to either continued treatment with aspirin 160 mg/d or change to clopidogrel 75mg/d after initial determination of their platelet reactivity while on aspirin treatment. Clinical endpoints will be recorded for at least 2 years and related to the initial aspirin response.

Scand Cardiovasc J. 2004 Dec;38(6):353-6.

ELIGIBILITY:
Inclusion Criteria:

* Stable, symptomatic coronary heart disease, verified by coronary angiography, being treated with angioplasty/stent implantation (PCI) or not.

Exclusion Criteria:

* Indication for warfarin treatment.
* Indication for or contraindication to the study drugs.
* Pregnancy or breast-feeding.
* Malignancy that may interfere with life expectancy.
* Psychiatric disease, mental retardation, dementia, drug abuse, alcoholism or conditions that can severely reduce compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2003-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 years
Myocardial infarction | 2 years
Unstable angina with ECG changes or raised levels of cardiac markers not to be classified as a myocardial infarction | 2 years

SECONDARY OUTCOMES:
Instent restenosis and/or thrombosis detected by coronary angiography. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alf-Aage R. Pettersen, M.D., Principal Investigator — Dept. of Cardiology, Ullevaal University Hospital, Oslo; Harald Arnesen, M.D. Ph.D., Study Chair — Center for Clinical Cardiovascular Research, Ullevaal University Hospital, Oslo; Ingebjorg Seljeflot, Ph.D., Study Director — Center for Clinical Cardiovascular Research, Ullevaal University Hospital, Oslo; Michael Abdelnoor, Ph.D., Study Director — Center for Clinical Cardiovascular Research, Ullevaal University Hospital, Oslo; Arne Westheim, M.D. Ph.D, Study Director — Dept. of Cardiology, Ullevaal University Hospital, Oslo
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Buchanan MR, Brister SJ. Individual variation in the effects of ASA on platelet function: implications for the use of ASA clinically. Can J Cardiol. 1995 Mar;11(3):221-7. PMID 7889440
- [Background] Grotemeyer KH. Effects of acetylsalicylic acid in stroke patients. Evidence of nonresponders in a subpopulation of treated patients. Thromb Res. 1991 Sep 15;63(6):587-93. doi: 10.1016/0049-3848(91)90085-b. PMID 1780803
- [Background] Gum PA, Kottke-Marchant K, Poggio ED, Gurm H, Welsh PA, Brooks L, Sapp SK, Topol EJ. Profile and prevalence of aspirin resistance in patients with cardiovascular disease. Am J Cardiol. 2001 Aug 1;88(3):230-5. doi: 10.1016/s0002-9149(01)01631-9. PMID 11472699
- [Background] Helgason CM, Bolin KM, Hoff JA, Winkler SR, Mangat A, Tortorice KL, Brace LD. Development of aspirin resistance in persons with previous ischemic stroke. Stroke. 1994 Dec;25(12):2331-6. doi: 10.1161/01.str.25.12.2331. PMID 7974569
- [Background] Hurlen M, Seljeflot I, Arnesen H. The effect of different antithrombotic regimens on platelet aggregation after myocardial infarction. Scand Cardiovasc J. 1998;32(4):233-7. doi: 10.1080/14017439850140021. PMID 9802142
- [Background] De Gaetano G, Cerletti C. Aspirin resistance: a revival of platelet aggregation tests? J Thromb Haemost. 2003 Sep;1(9):2048-50. doi: 10.1046/j.1538-7836.2003.00354.x. No abstract available. PMID 12941050
- [Background] Patrono C. Aspirin resistance: definition, mechanisms and clinical read-outs. J Thromb Haemost. 2003 Aug;1(8):1710-3. doi: 10.1046/j.1538-7836.2003.00284.x. No abstract available. PMID 12911581
- [Background] Grotemeyer KH, Scharafinski HW, Husstedt IW. Two-year follow-up of aspirin responder and aspirin non responder. A pilot-study including 180 post-stroke patients. Thromb Res. 1993 Sep 1;71(5):397-403. doi: 10.1016/0049-3848(93)90164-j. PMID 8236166
- [Background] Buchanan MR, Schwartz L, Bourassa M, Brister SJ, Peniston CM; BRAT Investigators. Results of the BRAT study--a pilot study investigating the possible significance of ASA nonresponsiveness on the benefits and risks of ASA on thrombosis in patients undergoing coronary artery bypass surgery. Can J Cardiol. 2000 Nov;16(11):1385-90. PMID 11109035
- [Background] Gum PA, Kottke-Marchant K, Welsh PA, White J, Topol EJ. A prospective, blinded determination of the natural history of aspirin resistance among stable patients with cardiovascular disease. J Am Coll Cardiol. 2003 Mar 19;41(6):961-5. doi: 10.1016/s0735-1097(02)03014-0. PMID 12651041
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Background] Hurlen M, Abdelnoor M, Smith P, Erikssen J, Arnesen H. Warfarin, aspirin, or both after myocardial infarction. N Engl J Med. 2002 Sep 26;347(13):969-74. doi: 10.1056/NEJMoa020496. PMID 12324552
- [Background] Andersen K, Hurlen M, Arnesen H, Seljeflot I. Aspirin non-responsiveness as measured by PFA-100 in patients with coronary artery disease. Thromb Res. 2002 Oct 1;108(1):37-42. doi: 10.1016/s0049-3848(02)00405-x. PMID 12586130
- [Background] Pettersen AA, Seljeflot I, Abdelnoor M, Arnesen H. Unstable angina, stroke, myocardial infarction and death in aspirin non-responders. A prospective, randomized trial. The ASCET (ASpirin non-responsiveness and Clopidogrel Endpoint Trial) design. Scand Cardiovasc J. 2004 Dec;38(6):353-6. doi: 10.1080/14017430410024324. PMID 15804802
- [Derived] Opstad TB, Nordeng J, Pettersen AR, Akra S, Bratseth V, Zaidi H, Helseth R, Solheim S, Seljeflot I. The NLRP3 Genetic Variant (rs10754555) Reduces the Risk of Adverse Outcome in Middle-Aged Patients with Chronic Coronary Syndrome. J Immunol Res. 2022 Dec 20;2022:2366695. doi: 10.1155/2022/2366695. eCollection 2022. PMID 36582742
- [Derived] Warlo EMK, Bratseth V, Pettersen AR, Holme PA, Arnesen H, Seljeflot I, Opstad TB. Genetic Variation in ADAMTS13 is Related to VWF Levels, Atrial Fibrillation and Cerebral Ischemic Events. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296221141893. doi: 10.1177/10760296221141893. PMID 36474435
- [Derived] Warlo EMK, Pettersen AR, Arnesen H, Seljeflot I. vWF/ADAMTS13 is associated with on-aspirin residual platelet reactivity and clinical outcome in patients with stable coronary artery disease. Thromb J. 2017 Nov 22;15:28. doi: 10.1186/s12959-017-0151-3. eCollection 2017. PMID 29200971
- [Derived] Pettersen AA, Seljeflot I, Abdelnoor M, Arnesen H. High On-Aspirin Platelet Reactivity and Clinical Outcome in Patients With Stable Coronary Artery Disease: Results From ASCET (Aspirin Nonresponsiveness and Clopidogrel Endpoint Trial). J Am Heart Assoc. 2012 Jun;1(3):e000703. doi: 10.1161/JAHA.112.000703. Epub 2012 Jun 22. PMID 23130135
- [Derived] Bratseth V, Pettersen AA, Opstad TB, Arnesen H, Seljeflot I. Markers of hypercoagulability in CAD patients. Effects of single aspirin and clopidogrel treatment. Thromb J. 2012 Aug 10;10(1):12. doi: 10.1186/1477-9560-10-12. PMID 22883224
- [Derived] Opstad TB, Pettersen AA, Arnesen H, Seljeflot I. Circulating levels of IL-18 are significantly influenced by the IL-18 +183 A/G polymorphism in coronary artery disease patients with diabetes type 2 and the metabolic syndrome: an observational study. Cardiovasc Diabetol. 2011 Dec 5;10:110. doi: 10.1186/1475-2840-10-110. PMID 22141572
- [Derived] Pettersen AA, Arnesen H, Opstad TB, Seljeflot I. The influence of CYP 2C19*2 polymorphism on platelet function testing during single antiplatelet treatment with clopidogrel. Thromb J. 2011 Mar 22;9:4. doi: 10.1186/1477-9560-9-4. PMID 21426546